CLINICAL TRIAL: NCT06407102
Title: Collection of Primary Human Nasal Epithelial Cells
Brief Title: Collection of Primary Human
Acronym: BIONOSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DR230317
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Nasal Disease
Keywords: nasal cells; Respiratory epithelium
MeSH Terms: conditions — Nose Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with programmed surgery (Other): Patient programmed with surgery of meatotomy, septoplasty or turbinoplasty, or other programmed surgeries
  Interventions: Other: Collection of nasal cells during programme surgery

INTERVENTIONS:
Other: Collection of nasal cells during programme surgery — During programmed surgery (meatotomy, septoplasty or turbinoplasty for example, or other programmed surgeries), the surgeon will take an atraumatic sample from the nasal cavity using a dedicated device (brush) from the healthy nasal mucosa.

SUMMARY:
Treatment and prevention of respiratory infections are of great interest in many medical areas. Create a physical device covered by primary human nasal cells could be very usefull in order to analyse delivery and efficiency of drugs. In this context the aim of this project is to create a collection of primary cells from the human nasal epithelium.

This collection will be realised during programmed surgery, thanks to a specific device dedicated to collect nasal cells. Then the cells will be sent to the lab in order to grow at the air-liquid interface, which is an excellent 'ex vivo' model for their study.

DETAILED DESCRIPTION:
The treatment and prevention of respiratory infections caused by emerging viruses or antibiotic-resistant bacteria are major societal and medical challenges. Inhalation allows drugs to be administered in the form of a spray or aerosol, directly into the respiratory tract (nose or lung). This is a validated approach for the non-invasive delivery of drugs to prevent and treat respiratory diseases, particularly infectious ones. Primary human nasal cell cultures grown at the air-liquid interface are an excellent 'ex vivo' model for their study in a physiological and pathophysiological context, and for testing new therapies, including aerosols. In addition, this culture model also offers an alternative to animal experimentation.

The aim of this project is therefore to create a collection of primary cells from the human nasal epithelium.

The main objective is to obtain a minimum of 60 samples of nasal epithelial cells from patients that can be cultured in air-liquid interface. The secondary objectives are to be able to study these nasal cells under physiological and pathophysiological conditions. The cells will first be amplified to constitute a cell biobank. They will then be studied under physiological conditions (anatomical and functional characterisation). Finally, they can be used to establish different models of infection or inflammation, in order to test future aerosol drugs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years) whose native language is French, or who understands French.
* Affiliation with a French social security system (CMU accepted).
* Informed consent, written and signed by the participant.
* Planned rhinological surgery (meatotomy, septoplasty or turbinoplasty for example, but other surgeries as well)

Exclusion Criteria:

* Patients under court protection, guardianship or curatorship.
* Pregnant or breast-feeding women (positive pregnancy test for women of childbearing age).
* Patients presenting a major alteration of the mucosa or a malignant rhinosinus pathology.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2027-05-02 (Estimated); Study Completion 2028-05-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of viability of nasal epithelial cells from the operating room to laboratory | 6 hours
  Collect nasal epithelial cells that can be grown in vitro in an air-liquid interface

SECONDARY OUTCOMES:
Percentage of efficacy of the procedure | 3 years
  Percentage of samples that can actually be cultivated following transfer to the laboratory.

IPD SHARING:
Plan to Share IPD: Undecided